CLINICAL TRIAL: NCT00865111
Title: A Randomized, Single Dose Two -Way Crossover Relative Bioavailability Study of Bupropion Sustained Release Tablets in Fasted, Normal, Healthy Men.
Brief Title: A Relative Bioavailability Study of Bupropion Sustained Release 150 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 06-0646-001
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Bupropion; Healthy subjects
MeSH Terms: interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Bupropion 150 mg Extended-Released Tablet, single dose
  Interventions: Drug: Bupropion 150 mg Extended-Released Tablet, single dose
- B (Active Comparator): Wellbutrin SR® 150 mg Sustained-Release Tablet, single dose
  Interventions: Drug: Wellbutrin SR® 150 mg Sustained-Release Tablet, single dose

INTERVENTIONS:
Drug: Bupropion 150 mg Extended-Released Tablet, single dose — A: Experimental Subjects received Abrika formulated products under fasting conditions
  Other Names: Bupropion
  Arms: A
Drug: Wellbutrin SR® 150 mg Sustained-Release Tablet, single dose — B: Active comparator Subjects received GlaxoSmithKline formulated products under fasting conditions
  Other Names: Bupropion
  Arms: B

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Abrika Bupropion 150 mg sustained release tablet to that of Wellbutrin SR sustained release tablet after a single, one-tablet dose in fasted subjects.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: A Randomized, Single Dose Two -Way Crossover Relative Bioavailability Study of Bupropion Sustained Release Tablets in Fasted, Normal, Healthy Men.

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man who volunteers to participate?
* Is he 18-45 years of age, inclusive?
* Is his BMI between 19 and 30, inclusive?
* Is he considered reliable and capable of understanding his responsibility and role in the study?
* Has he provided written informed consent? A no answer to any of the above questions indicates that the individual is ineligible for enrollment

Exclusion Criteria:

* Does the individual have a history of allergy or hypersensitivity to bupropion?
* Does he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his safety?
* Does he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, renal or other diseases, conditions or surgeries that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Does he have serious psychological illness?
* Does he have significant history (within the past year) or clinical evidence of alcohol or drug abuse?
* Does he have a positive urine drug screen or saliva alcohol screen, or a positive HIV-l, or hepatitis B or C screen?
* Has he consumed grapefruit or grapefruit juice during the 7-day period preceding study initiation?
* Is he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the last blood sample has been taken in each study period?
* Has he used any prescription drug during the 14-day period prior to study initiation, or any OTC drug during the 72-hour period preceding study initiation?
* Is he unable to refrain from the use of all concomitant medications during the study?
* Has he donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?
* Has he donated plasma during the two week period preceding study initiation?
* Has he received an investigational drug during the 30 day period preceding study initiation?
* Is he a heavy smoker (usually smoking more than 25 cigarettes per day? A yes answer to any of the above questions indicates that the individual is ineligible for enrollment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R. Pizarro,, M.D., Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC Ft. Myers, Inc., Fort Myers, Florida, United States